CLINICAL TRIAL: NCT04702503
Title: A Phase 1b Study Evaluating the Safety and Efficacy of Topical Administration of WP1220, an Inhibitor of STAT3 Activation, in Adults With Stage I, II, or III Mycosis Fungoides (Cutaneous T-Cell Lymphoma, CTCL)
Brief Title: Study of WP1220 for the Treatment of Adult Subjects With Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Moleculin Biotech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MB-201
Record Dates: First submitted 2019-03-19; First posted 2021-01-11 (Actual); Last update posted 2021-01-11 (Actual); Status verified 2021-01

CONDITIONS: Cutaneous T-Cell Lymphoma/Mycosis Fungoides
MeSH Terms: conditions — Mycosis Fungoides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10% WP1220 ointment (Experimental): 10% WP1220 ointment topically applied 2x day for 84 days
  Interventions: Drug: WP1220

INTERVENTIONS:
Drug: WP1220 — Topical administration 2x daily for 84 consecutive days

SUMMARY:
Single center, pilot study to evaluate the safety and efficacy topical administration of WP1220 in subjects with Stage I, II or III Mycosis Fungoides (CTCL)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at the time of signing informed consent.
2. Clinical diagnosis of MF.
3. Stage IA, IB, IIA, IIB, or II MF: T1-T4 with measurable lesions
4. Previously treatment with at least one standard therapy used to treat Stage IA, IB, IIA, IIB, or III MF.
5. Measurable skin disease must have at least 2 eligible baseline index lesions with maximum total area ≤ 40 cm2. Eligible lesions must be below the head (face and scalp are excluded) and must not involve the genitalia or anus.
6. ECOG performance status of 0-2
7. Subject must read and sign informed consent form and be willing to comply with the instructions, restrictions, nature and procedures of the study.
8. Willing to avoid tanning devices or exposure of the treated skin to the sun.
9. Willing to not use cosmetics, including lotions, creams, and moisturizers on the treated lesions.
10. Willing to use topical steroid on a maximum of 25% of BSA occupied by MF on areas not involved in the clinical trial.
11. Must have recovered from the effects of surgery requiring general anesthesia and intubation for a minimum of 3 months, and from minor surgery requiring only local anesthetic for a minimum of 2 weeks.
12. Concomitant disease must be stable and subjects must be on the same dose and schedule of any medications for at least 1 month before screening.
13. Subjects of both genders who are of childbearing potential including perimenopausal women who are fewer than 2 years from their last menses, must use one of the following effective means of contraceptionL

    * Birth control pills in conjunction with spermicide gel
    * Surgical sterilization
    * Intra uterine device
    * Condom and spermicide gel together
    * Sexual abstinence during study period

The requirements above do not apply to:

* Postmenopausal women with spontaneous amenorrhea for at least 2 years, or
* Subjects with bilateral oophoerctomy with or without a hysterectomy and an absence of bleeding for at least 6 months, or
* Subjects with total hysterectomy and an absence of bleeding for at least 3 months

Exclusion Criteria:

1. MF with no prior therapy.
2. Subjects with a diagnosis of stage IV MF at Screening or subsequently observed at Baseline.
3. Subjects with unusual phenotypes, e.g. lymphomatoid papulosis MF-like type.
4. Subjects who require immediate treatment for progressive MF.
5. Subjects treated with at least one of the following methods within 8 weeks prior to

   Baseline:
   * Total body electron beam radiation
   * Investigational drugs or treatments
6. Subjects treated with at least one of the following methods within 4 weeks prior to

   Baseline:
   * Local radiation therapy
   * UVB therapy
   * PUVA
   * Topical chemotherapy
   * Topical corticosteroids or retinoids
   * Systemic chemotherapeutic agents (excluding low doses of MTX max. 25 mg/wk)
7. Index lesion treatment with at least one of the following methods within 2 weeks prior to Baseline:

   * Any surgical procedures other than biopsies related to CTCL diagnosis or follow- up
   * Any topical treatment other than bland moisturizers (creams, lotions, emollients, etc)
8. Skin infections on screening or baseline involving index lesions planned to be treated in the clinical trial.
9. The presence of any clinically significant laboratory abnormalities at screening including, but not limited to abnormalities of the white blood count, hemoglobin, platelets, serum chemistry (glucose, uric acid, calcium, phosphorus, sodium, potassium, chloride, alkaline phosphatase, albumin and total bilirubin), thyroid stimulating hormone, fT3 and fT4 as determined by the Investigator in conjunction with the Medical Monitor.
10. Any significant uncontrolled medical disease as evaluated by the Investigator and/or Medical Monitor, chronic or active within the past 6 months, including but not limited to, cardiac disease, seizure disorder, liver disease, renal disease, chronic infection, uncontrolled diabetes, lung disease.
11. Any prior history or active malignancy other than MF.
12. Subjects in deep depression.
13. Subjects who are not mentally capable of understanding the protocol and all procedures.
14. Subjects who do not agree to have the necessary blood draws and procedures for laboratory tests and evaluations according to protocol.
15. Known allergy to any active or inactive ointment ingredient.
16. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-11-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the safety profile of WP1220 applied topically (adverse events) | 12 weeks (3 28-day cycles)
  Safety will be evaluated by reported adverse events

SECONDARY OUTCOMES:
Evaluation of WP1220 applied topically to index lesions via standard measurement scale | 12 weeks
  Efficacy to be demonstrated through ≥50% improvement in standard assessments of lesions in comparison to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Silberman, MD, PhD, Study Director — Moleculin Biotech, Inc.
Locations (1):
- Medical University of Gdansk, Gdansk, Poland